CLINICAL TRIAL: NCT07059767
Title: A Phase IIa, Double-blind, Randomized, Placebo-controlled Trial in Participants With Asthma to Evaluate the Impact of Intranasal ETH47 on the Development of Asthma-related Symptoms Following Rhinovirus Challenge
Brief Title: Phase IIa Trial in Participants With Asthma to Evaluate Impact of Intranasal ETH47 on Development of Asthma-related Symptoms Following Rhinovirus Challenge
Acronym: ETH47-201
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ethris GmbH (Industry)
Collaborators: VirTus Respiratory Research Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ETH47-201; ISRCTN21576805 (Other: ISRCTN)
Record Dates: First submitted 2025-06-27; First posted 2025-07-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Asthma (Diagnosis)
MeSH Terms: conditions — Asthma; Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ETH47 (Experimental)
  Interventions: Drug: ETH47
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ETH47 — single intranasal dose of ETH47
  Arms: ETH47
Drug: Placebo — single intranasal dose of placebo
  Arms: Placebo

SUMMARY:
A Phase IIa trial in participants with asthma to evaluate the impact of intranasal ETH47 on the development of asthma-related symptoms following rhinovirus challenge

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Participants aged ≥18 and ≤65 years at the time of obtaining informed consent.
3. Diagnosis of clinical asthma (>12% reversibility following short acting beta 2 agonist (SABA) treatment or PC20 methacholine challenge of <8 mg/mL).
4. Stable (no change in medication or dose) asthma maintenance therapy with inhaled glucocorticosteroids (ICS) or ICS + long acting beta 2 agonist (LABA) for at least 3 months prior to dosing.
5. Clinically stable with no exacerbations within 3 months prior to dosing.
6. Sero-negative test result to RV-A16.
7. Participants must agree to use contraception methods (if applicable).

Exclusion Criteria:

1. Any cold symptom within the last month such as sore throat, sneezing, rhinorrhoea, malaise, nasal obstruction or cough.
2. Evidence of current allergic rhinitis, including perennial allergic rhinitis, or rhinosinusitis or nasal polyps.
3. History of or current diagnosis of chronic obstructive pulmonary disease, emphysema, cystic fibrosis or bronchiectasis.
4. The evidence of any other historic, active or chronic disease following a detailed medical and surgical history which, in the Investigator's judgement, puts the participant at risk due to participation in the trial, may influence the results of the trial, or the participant's ability to participate in the trial. This includes a history of emergency room visits or hospital admissions due to common cold.
5. Current vaper or smoker, or ex-smoker who stopped within the last 12 months or with a >5 year pack history; current vapers may be included if willing to stop prior to Baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in peak of total lower respiratory symptoms score (LRSS) | Day 1 to Day 14
  7 Questions on lower respiratory symptoms are scored from 0-3 (absent, mild moderate, severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Virtus Respiratory Research Ltd and Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No